CLINICAL TRIAL: NCT05035745
Title: Phase I Dose Finding Study of Selinexor and Talazoparib in Patients With Advanced Refractory Solid Tumors, Followed by Phase II Expansion Cohort Study in Patients With Advanced/ Metastatic Triple Negative Breast Cancers. (START)
Brief Title: Selinexor & Talazoparib in Advanced Refractory Solid Tumors; Advanced/Metastatic Triple Negative Breast Cancer (START)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC01/05/20; IST-325 (KPT)
Record Dates: First submitted 2021-03-01; First posted 2021-09-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Advanced Refractory Solid Tumors; Advanced Triple Negative Breast Cancers; Metastatic Triple Negative Breast Cancers
Keywords: Selinexor; Talazoparib; breast cancer; Triple negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — talazoparib; selinexor

STUDY DESIGN:
Intervention Model Description: Phase I Patients will be treated with Talazoparib daily and Selinexor once per week (3 out of 4 weeks), on a 4 weekly cycle (28 days) in a modified 3+3 dose escalation/ de-escalation design
  Phase II Patients with advanced/ metastatic triple negative breast cancer, unselected for known platinum sensitivity or resistance, will be enrolled. A pilot of 10 patients will be enrolled. If 0-1 patients achieve an objective response, the combination is deemed to be of no interest for further development. If 2 or more of 10 patients achieve an objective response, another 20 patients will be enrolled to confirm the objective response rate. In the final objective response analysis, TNBC patients will be stratified into platinum-naïve/platinum sensitive versus platinum-resistant to determine if prior platinum sensitivity impacts objective response rates to the combination of Talazoparib and Selinexor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with refractory solid tumors (Experimental): Phase I will be carried out in a modified 3+3 dose escalation design, with a projected enrolment of patients with refractory solid tumors to determine the RP2D.
  Interventions: Drug: Talazoparib; Drug: Selinexor

INTERVENTIONS:
Drug: Talazoparib — Patients will be treated with Talazoparib daily on a 4 weekly cycle (28 days)
Drug: Selinexor — Patients will be treated with Selinexor once per week (3 out of 4 weeks), on a 4 weekly cycle (28 days)

SUMMARY:
This is a single arm, open-label, phase I dose finding study, followed by a phase II expansion study. Phase I will be carried out in a modified 3+3 dose escalation design, with a projected enrolment of 33 patients with refractory solid tumors to determine the RP2D. In the phase II portion, a total of 30 patients with advanced/metastatic TNBC will be enrolled.

DETAILED DESCRIPTION:
Hypothesis The investigators hypothesize that the combination of Talazoparib and Selinexor will have clinical efficacy in TNBC, independent of BRCA mutation status.

Primary Objectives

* To determine the safety profile of combination of Talazoparib and Selinexor in advanced/ metastatic solid tumors.
* To determine the RP2D of Talazoparib and Selinexor combination therapy in patients with advanced/ metastatic solid tumors.

Secondary Objectives

• To determine the objective response rate to combination Talazoparib and Selinexor in advanced/ metastatic TNBCs.

Exploratory Objectives

* To assess the effect of the combination on pharmacokinetics of Talazoparib and Selinexor
* To explore the impact of pharmacogenetics on toxicity and efficacy of combination Talazoparib and Selinexor.
* To assess changes in circulating tumor cells and plasma biomarkers during treatment.
* To assess pharmacodynamic changes and predictive biomarkers in tumor tissue during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent in accordance with local institutional guidelines.
2. All patient must not have received prior PARPi including talazoparib
3. All patients must not have prior therapy with selinexor.
4. Age ≥ 18
5. Estimated life expectancy of at least 12 weeks.
6. Has recovered from acute toxicities from prior anti-cancer therapies to grade 2 or lower.
7. a) Dose escalation phase: Patients with histologically or cytologically confirmed advanced or metastatic solid tumors who have radiological evidence of progressive disease on study entry that is deemed unlikely to benefit from further conventional therapy, or for which no standard therapy is available.

   b) Dose expansion phase: Patients with previously treated, advanced or metastatic histologically or cytologically confirmed triple negative breast cancers. Patients must have evidence of progressive disease on study entry after at least one line of anti-cancer therapy. Patients will be stratified into platinum-naïve (not having been treated with platinums-containing chemotherapy in the neoadjuvant, adjuvant or palliative setting), platinum sensitive (defined as having prior objective response or sustained disease control lasting ≥6 months to platinum-containing chemotherapy in the metastatic setting, or relapsed ≥6 months after completing neoadjuvant or adjuvant platinums-containing chemotherapy), and platinum resistant (defined as having progressive disease as the best response or disease control <6 months to platinum-containing chemotherapy in the metastatic setting, or relapsed <6 months after completing neoadjuvant or adjuvant platinums-containing chemotherapy).

   There is no upper limit on the number of prior treatments provided all inclusion/exclusion criteria are met. Hormone ablation therapy is considered an anti-cancer regimen. Radiation and surgery are not considered anti-cancer regimens.
8. Measurable disease by RECIST 1.1 criteria.
9. Eastern cooperative Oncology Group (ECOG) Performance Status of 0-1
10. Adequate bone marrow function and organ function within 2 weeks of study treatment

    1. Adequate hematologic function defined as:

       * Absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L
       * Platelets ≥ 125 x 109/L during dose escalation phase; platelets ≥ 100 x 109/L during dose expansion phase
       * Hemoglobin ≥ 9 x 109/L
    2. Hepatic function:

       * Bilirubin ≤ 1.5 times the upper limit of normal (ULN)
       * ALT or AST ≤ 2.5 times ULN (or ≤ 5 times ULN with liver metastases)
    3. Adequate renal function:

       * Calculated creatinine clearance of ≥ 60 mL/min, calculated using the formula of Cockroft and Gault: (140-Age) x Mass (kg)/(72 x creatinine mg/dL); multiply by 0.85 if female.
11. Able to swallow tablets/ pills.
12. Able to comply with study-related procedures.
13. Female patients of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective methods of contraception throughout the study and for 7 months following the last dose of study treatment

Exclusion Criteria:

1. Treatment within the last 30 days with any investigational drug.
2. Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy
3. Major surgery within 28 days of study drug administration
4. Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
5. Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
6. Pregnancy
7. Breast feeding
8. Poorly controlled diabetes mellitus
9. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment (for phase II only).
10. Symptomatic brain metastasis.
11. History of significant neurological or mental disorder, including seizures or dementia.
12. Unable to comply with study procedures
13. Current or anticipated use of strong P-gp inhibitors: amiodarone, carvedilol, clarithromycin, cobicistat, darunavir, dronedarone, erythromycin, indinavir, itraconazole, ketoconazole, lapatinib, lopinavir, propafenone, quinidine, ranolazine, ritonavir, saquinavir, telaprevir, tipranavir, valspodar, verapamil
14. Current or anticipated use of strong BCRP inhibitors: curcumin, cyclosporine A, eltrombopag, elacridar, fumitremorgin C, novobiocin, sulfasalazine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
safety profile of combination of Talazoparib and Selinexor in advanced/ metastatic solid tumors using NCI CTCAE toxicity grading version 5.0. | 5 years
  Patients with advanced/ metastatic triple negative breast cancer, unselected for known platinum sensitivity or resistance, will be enrolled. A pilot of 10 patients will be enrolled. If 0-1 patients achieve an objective response, the combination is deemed to be of no interest for further development. If 2 or more of 10 patients achieve an objective response, another 20 patients will be enrolled to confirm the objective response rate. In the final Safety evaluations will be performed for all patients prior to each cycle of treatment, and include taking a medical history, physical examination, adverse event documentation, full blood count, renal function, liver function tests and electrocardiogram (ECG).
  Toxicities will be graded using the NCI CTCAE toxicity grading version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmid P, Adams S, Rugo HS, Schneeweiss A, Barrios CH, Iwata H, Dieras V, Hegg R, Im SA, Shaw Wright G, Henschel V, Molinero L, Chui SY, Funke R, Husain A, Winer EP, Loi S, Emens LA; IMpassion130 Trial Investigators. Atezolizumab and Nab-Paclitaxel in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2018 Nov 29;379(22):2108-2121. doi: 10.1056/NEJMoa1809615. Epub 2018 Oct 20. PMID 30345906
- [Background] Robson ME, Tung N, Conte P, Im SA, Senkus E, Xu B, Masuda N, Delaloge S, Li W, Armstrong A, Wu W, Goessl C, Runswick S, Domchek SM. OlympiAD final overall survival and tolerability results: Olaparib versus chemotherapy treatment of physician's choice in patients with a germline BRCA mutation and HER2-negative metastatic breast cancer. Ann Oncol. 2019 Apr 1;30(4):558-566. doi: 10.1093/annonc/mdz012. PMID 30689707